CLINICAL TRIAL: NCT03799861
Title: Newborn Heart Rate as a Catalyst for Improved Survival (NeoBeat Study)
Brief Title: Newborn Heart Rate as a Catalyst for Improved Survival
Status: Completed | Type: Observational
Sponsor: American Academy of Pediatrics (Other)
Collaborators: Kinshasa School of Public Health (Other); Laerdal Global Health (Other); RTI International (Other); Thrasher Research Fund (Other); University of North Carolina, Chapel Hill (Other); Saving Lives at Birth (Unknown)
Responsible Party: Sponsor
Other Study IDs: 7200AA18FA00010
Record Dates: First submitted 2018-11-09; First posted 2019-01-10 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Stillbirth; Neonatal Respiratory Depression; Neonatal Bradycardia; Neonatal Resuscitation
Keywords: Neonatal Resuscitation; Stillbirth; Neonatal Respiratory Depression; Neonatal Bradycardia
MeSH Terms: conditions — Stillbirth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Epoch 1: Care prior to HBB training: A period of demographic and birth outcome data collection for a retrospective cohort of all infants born in the three study hospitals during the 18 months prior to the start of Epoch 2, reflecting care prior to HBB training.
- Epoch 2: HBB with NeoBeat: Implementation of Helping Babies Breathe training in combination with NeoBeat for detection of HR in non-breathing newborns, after which demographic and birth outcome data will be abstracted from the medical record along with observational data on resuscitation for prospective cohort of all infants born in the three study hospitals for a 9-month period.
  Interventions: Other: Epoch 2: HBB with NeoBeat
- Epoch 3: HR-guided HBB: Implementation of HR-guided Helping Babies Breathe training with NeoBeat for measurement of HR throughout resuscitation of non-breathing newborns, after which demographic and birth outcome data will be abstracted from the medical record along with observational data on resuscitation for a prospective cohort of all infants born in the three study hospitals for a 9-month period.
  Interventions: Other: Epoch 3: HR-guided HBB

INTERVENTIONS:
Other: Epoch 2: HBB with NeoBeat — At the beginning of Epoch 2, all birth attendants in each of the 3 maternity units will participate in a 2 day workshop in Kinshasa in French that will include instructions regarding use of NeoBeat and training in HBB 2.0. Participants will be introduced to NeoBeat, which will include practice with NeoBeat using the NeoNatalie newborn simulator. This training will be conducted in French using typical adapted training materials for this program that incorporate placement of NeoBeat at appropriate times in the algorithm, including a flipchart and NeoNatalie. Participants will complete the pre and post knowledge check questionnaire for the training as well as the Observed Standardized Clinical Exams (OSCEs) with the incorporation of use of NeoBeat into the OSCEs.
  Groups: Epoch 2: HBB with NeoBeat
Other: Epoch 3: HR-guided HBB — At the beginning of Epoch 3, all birth attendants in each of the 3 maternity units will participate in a 1 day workshop in Kinshasa in French that will instruct them in an adapted, HR-guided HBB algorithm. This training will include simulation with NeoNatalie and NeoBeat. Participants will complete a pre and post knowledge check questionnaire for the training as well as the Observed Standardized Clinical Exams (OSCEs).
  Groups: Epoch 3: HR-guided HBB

SUMMARY:
Heart rate (HR) is not routinely assessed during newborn resuscitations in low- and lower-middle income countries (LMICs). Many non-breathing newborns classified as fresh stillbirths have a heartbeat and are live born. The effect of a low-cost monitor for measuring HR on the problem of misclassification of stillbirths in LMICs is unknown.

Knowledge of HR during newborn resuscitation might also result in timely administration of appropriate interventions, and improvement in outcomes. Helping Babies Breathe (HBB), a resuscitation algorithm developed by the American Academy of Pediatrics (AAP), is widely accepted as the standard of care for newborn resuscitation in low-resource settings. In keeping with the International Liaison Committee on Resuscitation (ILCOR) recommendations that HR be measured during newborn resuscitation, HBB calls for HR assessment after 1 minute of positive-pressure ventilation with good chest movement (or sooner if there is a helper who can palpate/auscultate heart rate). However, given the frequent reality of a single provider attending deliveries in LMICs, as well as the currently available methods for assessing HR (i.e. palpitation or auscultation), assessment of HR is challenging to perform without delaying or stopping the provision of other life-saving interventions such as bag and mask ventilation. The effect of low-cost, continuous HR monitoring to guide resuscitation in these settings is unknown.

NeoBeat is a low-cost, battery-operated device designed by Laerdal Global Health for the measurement of newborn HR. The device can be placed rapidly on a newborn by a single provider, and within 5 seconds, displays HR digitally. A preliminary trial of NeoBeat in 349 non-breathing newborns in Tanzania detected a HR in 67% of newborns classified as stillbirths, suggesting up to two thirds of fresh stillbirths may be misclassified in similar settings.

This trial will evaluate: 1) the effectiveness of HBB in combination with NeoBeat for vital status detection on reduction of reported stillbirths, and 2) the effectiveness of HR-guided HBB on effective breathing at 3 minutes.

The primary hypothesis is that implementation of HBB with measurement of HR using NeoBeat will decrease the reported total stillbirth rate by 15% compared to standard care. The secondary hypothesis is that implementation of HR-guided HBB will increase the proportion of newborns not breathing well at birth who are effectively breathing at 3 minutes by 50% compared to HBB with NeoBeat.

ELIGIBILITY:
Inclusion Criteria: all newborns delivered via vaginal, assisted or operative delivery at any of 3 participating maternity units in Kinshasa, Democratic Republic of Congo (DRC), during the study period will be enrolled. All newborns will be included, regardless of:

* intrauterine fetal demise
* birth weight
* congenital anomalies
* multiple gestation
* any maternal complication

Exclusion Criteria:

* Newborns transferred to the maternity unit following delivery at a referral hospital or in the community
* Miscarriages, or previable newborns, defined as gestational age <28 weeks (or if gestational age is unavailable, birth weight <1,000g) at the time of delivery

Ages: 28 Weeks to 45 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All newborns delivered at any of the following 3 maternity units in Kinshasa, DRC over 3 years: Bumbu, Kingasani and Binza-Delvaux. The first 18 months of patients enrolled in the study will be retrospective, while the subsequent 18 months will be prospective. The entire study population will include non-observed and observed deliveries. Observed deliveries will be a convenience sample of non-breathing newborns based on availability of study nurses.
Sampling Method: Non-Probability Sample
Enrollment: 24034 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Reported Total Stillbirth Rate | At delivery
  The total number of stillborn infants (both fresh and macerated) at the facility per 1,000 births, with stillbirth as classified by the delivery attendant.

SECONDARY OUTCOMES:
Effective, Spontaneous Breathing at 3 Minutes | At 3 minutes of life
  Breathing without the assistance of stimulation or bag and mask ventilation at a respiratory rate ≥ 40 breaths per minute with a HR ≥ 100 beats per minute at 32 minutes of life.

OTHER OUTCOMES:
Fresh Stillbirth Rate | At delivery
  Total number of non-breathing newborns without a HR at the time of birth, and without signs of maceration, as determined by the delivery attendant, per 1,000 births.
Macerated Stillbirth Rate | At delivery
  Total number of non-breathing newborns without a HR at the time of birth, with signs of maceration, as determined by the delivery attendant, per 1,000 births.
Neonatal Death Prior to Discharge | Up to 28 days of life
  Death of a live born infant during the birth hospitalization, where death occurs prior to discharge or transfer from the facility of birth.
Number of Providers Adhering to Resuscitation Algorithm | At delivery
  any number of provider actions to promote resuscitation of the non-breathing newborn such as suctioning, stimulation, bag and mask ventilation and corrective measures to improve bag and mask ventilation in response to newborn respiratory condition or HR as defined in the resuscitation algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Bose, MD, Study Director — University of North Carolina, Chapel Hill; Jackie Patterson, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill; Sara Berkelhamer, MD, Study Chair — University at Buffalo; Nalini Singhal, MD, Study Chair — University of Calgary
Locations (3):
- Democratic Republic of the Congo (3):
  - Binza-Delvaux Maternity Hospital, Kinshasa
  - Centre Hospital Kingasani, Kinshasa
  - Mother and Child Hospital Bumbu, Kinshasa

IPD SHARING:
Plan to Share IPD: Yes